CLINICAL TRIAL: NCT04670029
Title: Impact of an Adapted Physical Activity Program on Event-free Survival in Patients With Diffuse Large-cell B Lymphoma Treated in 1st Line
Brief Title: Impact of an APA Program on EFS in Patients With Diffuse Large-cell B Lymphoma Treated in 1st Line
Acronym: PHARAOM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Weprom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WP-2020-03; 2019-A02248-49 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-04

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (No Intervention)
- APA (Experimental): * During the first 3 cures, 3 APA sessions will be offered per week:
    * 2 sessions of anaerobic type of 1 hour with muscle strengthening, stretching, flexibility and balance, supervised in the room,
    * 1 aerobic type exercise session of 1.5 hours (Nordic walking: outdoors) or a 3rd indoor session if not possible,
    * + home exercise book if the patient so wishes with record the time in minutes per session and the intensity felt and the modalities of the exercises carried out.
  * During the 5 remaining cycles, 3 APA sessions will be offered per week:
    * 1 session of 1 hour in an anaerobic exercise room (muscle strengthening, stretching, flexibility, balance) supervised,
    * 1 session of anaerobic exercise per week in autonomy at home (with exercise book),
    * 1 or more session per week of one hour of walking or cycling independently at home (aerobic effort) with declaration in the logbook of the intensity of exertion felt and the time in minutes per session.
  Interventions: Other: Adapted physical activity

INTERVENTIONS:
Other: Adapted physical activity — APA sessions during chemotherapy with aerobic and anaerobic sessions on site and at home (+ home exercises book if the patient so wishes)
  Arms: APA

SUMMARY:
Diffuse large B cell lymphoma is the most common histology of non-Hodgkin's malignant lymphomas (31% of lymphomas), with an incidence of between 15 and 20 new cases per year per 100,000 inhabitants in France. The median age is 65 and a third of patients are over 75 years old. 60% of patients are cured after a standard regimen of chemotherapy with RCHOP; 40% of patients will, however, relapse. No other regimen has shown improvement in overall survival, but poor prognosis factors have been identified. Beyond these factors, other prognostic factors can impact overall and progression-free survival: sarcopenia, nutritional status disorders Sarcopenia is defined by the reduction of muscle mass and strength. It was first described in the elderly and classified as geriatric syndrome such as dementia, falls or frailty. It varies from 5 to 13% between 60 and 70 years and between 11 and 50% beyond 80 years and is classified as primitive, that is to say related to age It can however be secondary to neoplasia. This event has been described in patients with hematologic malignancies during chemotherapy and can reach 55% of patients in the elderly. It is proportional to the intensity of the treatments. It emerges as an independent prognostic factor which is detrimental to survival in these patients. Physical exercise combined with nutritional support could reduce it.

The positive impact of adapted physical activity has been shown in numerous publications on reducing the incidence and risk of relapse for certain cancers (breast, colon prostate). It is less obvious in hematology in view of studies published on adapted physical activity . Adapted physical activity seems to provide a survival benefit in diffuse large cell B lymphoma however the number remains too low in this histology.

Sarcopenia is an often-underestimated event and is associated with older age, co-morbidities, increased infectious complications, and early mortality.

Correcting sarcopenia through appropriate physical activity could reduce its negative prognostic impact.

The aim of the study is to increase the event-free survival of patients in the RCHOP and adapted physical activity arm by 15% compared to the standard arm.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with diffuse large-cell B lymphoma regardless of the WHO 2016 classification subtype, or low-grade B lymphoma immediately transformed into high-grade B lymphoma (follicular lymphoma of the marginal zone, MALT, lymphocytic, lympho-plasma cells),
2. Treatment naïve or having benefited from 2 cycles of chemotherapy (prephase or COP and cycle n ° 1 of RCHOP) if Performance Status> 3 linked to hemopathy and reversible (≤ 2)
3. Aged ≥ 65 years old,
4. Eligible for treatment with RCHOP, regardless of the IPI score adjusted for age,
5. Performance Status ≤ 2,
6. Patient affiliated to a social security scheme,
7. Patient who has given written consent before any specific procedure related to the study

Exclusion Criteria:

1. Any other type of lymphoma (T lymphoma, Burkitt's lymphoma, non-transformed low-grade B lymphoma, etc.),
2. Cerebral or meningeal damage related to hemopathy,
3. Acquired or congenital motor or sensory deficit which does not allow the completion of APA sessions,
4. Uncontrolled arterial hypertension,
5. Disabling heart or respiratory failure not allowing the completion of APA sessions,
6. Disabling osteo-articular or muscular pathology,
7. LVEF <50%,
8. Patient having received 3 or more cycles of 1st line chemotherapy,
9. Pregnancy or breastfeeding,
10. Active viral infection: hepatitis B, C and HIV,
11. Persons deprived of their liberty or under guardianship
12. Dementia, mental alteration or psychiatric pathology which could compromise the patient's informed consent and / or compliance with the protocol and follow-up of the trial,
13. Patient who can't follow protocol for psychological, social, family or geographic reasons

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
To detect an absolute difference of 15% in event-free survival between the 2 groups | 5 years
  Event-free survival will be defined as the time between the date of inclusion and the date of the event or the date of the latest news if the patient is censored.

SECONDARY OUTCOMES:
The compliance with the 72 sessions of APA | 6 months
  Number of sessions performed per patient per part of the program
The overall physical activity load per patient and per session | 6 months
  Evaluated according to the Foster method (duration of the session in minutes x perceived effort according to the modified Borg scale)
The overall survival | 5 years
  Time between the date of inclusion and the date of death if the patient is deceased or the date of the latest news if the patient is censored
The progression free survival | 5 years
  time between the inclusion date and the date of the first examination showing Progression of the disease or the date of death if the patient is deceased or the date of the latest news if the patient is censored
The progression-free survival after relapse and resumption of therapy | 5 years
  Time between the date of the start of re-treatment and the date of the first examination showing progression of the disease or the date of death if the patient has died or the date of the latest news if the patient is censored,
The complete and partial response rates | 1 year
  according to Lugano criteria
The prevalence of complications | 6 months
  Number of patients who presented complication in the numerator and the number of patients followed in the denominator
The incidence of sarcopenia during follow-up | 2 years
  by CT scan during follow-up will be evaluated by the number of patients with sarcopenia diagnosed during follow-up in the numerator and the number of patients followed in the denominator
The prevalence of nutritional disorders at diagnosis and at the end of treatment | 6 months
  The number of patients with a disorder of nutritional status in the numerator and the number of patients followed in the denominator,
The rate of endocrinopathies | 6 months
  Number of patients with endocrinopathy between the inclusion date and the study discharge date in the numerator and the number of patients followed in the denominator
The rate of second cancers | 5 years
  Number of patients who presented with a second cancer during the study
The rate of cardiovascular events | 5 years
  Number of patients with a cardiovascular event
The quality of life of patients | 5 years
  Change from baseline of the European Organisation for Research and Treatment of Cancer quality of life C30 questionnaire score (higher score means better outcome)
The fatigue of patient | 5 years
  Change from baseline of Multidimensional fatigue inventory score (higher score means worse outcome)
The depression of patient | 5 years
  Change from baseline of Geriatric depression scale (higher score means worse outcome)
The cost of hospitalizations | 5 years
  Hospitalizations will be quote (economic data) by medical information department of center

CONTACTS AND LOCATIONS:
Overall Officials: Katell LE DÛ, MD, Principal Investigator — Clinique Victor Hugo/Centre Jean Bernard
Locations (5):
- France (5):
  - CHU Jean Minjoz, Besançon
  - Clinique Victor Hugo / Centre Jean Bernard, Le Mans
  - CHRU Nancy, Nancy
  - Hôpital Privé du Confluent, Nantes
  - CH Perpignan, Perpignan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dubu J, Boyas S, Roland V, Landry S, Septans AL, Balavoine M, Bourgeois H, Pointreau Y, Denis F, Letellier C, Le Du K. Physical Activity Program for the Survival of Elderly Patients With Lymphoma: Study Protocol for Randomized Phase 3 Trial. JMIR Res Protoc. 2022 Nov 25;11(11):e40969. doi: 10.2196/40969. PMID 36427234